CLINICAL TRIAL: NCT02438592
Title: PHASES: Provision of HIV Treatment at ATN Sites: An Evaluation for Stakeholders
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 125
Record Dates: First submitted 2015-04-02; First posted 2015-05-08 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-03

CONDITIONS: HIV
Keywords: Continuum of care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational study involving retrospective and prospective medical record review covering a total maximum of 104 weeks (24 months) per subject. An Audio Computer- Assisted Self-Interview (ACASI) at study entry will assess demographic and psychosocial variables of study subjects. Data will also be collected to assess clinic level variables. Definitions of engagement, prescription of antiretroviral therapy (ART), and viral suppression in the Continuum of Care (CoC) will utilize common definitions including those by U.S. Department of Health and Human Services (DHHS) and Health Resources and Services Administration (HRSA) HIV/AIDS Bureau (HAB). Data will be collected in a large, simple trial design manner to provide all elements for both the primary and secondary outcomes.

DETAILED DESCRIPTION:
This is an observational study involving retrospective and prospective medical record review covering a total maximum of 104 weeks (24 months) per subject. Behavioral data will be collected via ACASI at study entry to assess demographic and psychosocial variables of study subjects. All other data (biomedical, ART, healthcare utilization) at subsequent study visits will be collected via medical record abstraction. Information about missed visits as well as other healthcare utilization data can be abstracted from electronic appointment systems or other electronic systems at the clinical sites. Subject data will be abstracted from medical records for up to a maximum 26 weeks prior to the baseline study visit, as well as up to a maximum 78 weeks after the baseline study visit or through January 31, 2017, whichever occurs first, for a total maximum of 104 weeks or two years per subject. Data will also be collected from each Adolescent Medicine Trials Unit to assess clinic level variables at baseline (within 30 days of protocol registration) and 48 and 96 weeks after baseline. Definitions of engagement, prescription of antiretroviral therapy (ART), and viral suppression in the Continuum of Care (CoC) will utilize common definitions including those by U.S. Department of Health and Human Services (DHHS) and Health Resources and Services Administration (HRSA) HIV/AIDS Bureau (HAB). Data will be collected in a large, simple trial design manner to provide all elements for both the primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory evidence of HIV-1 infection per Centers for Disease Control and Prevention (CDC) Surveillance Case Definition for HIV Infection, 2014 (Section 1.1) http://www.cdc.gov/mmwr/preview/mmwrhtml/rr6303a1.htm;
* Behaviorally-acquired HIV after age 9 years;
* Age 13 through 24 years, inclusive, at the baseline visit (Enrollment);
* Planning to receive HIV medical care at an AMTU or at any clinical site that is part of the AMTU for the duration of study follow-up

  • If transition to an adult health care provider must occur during the course of study participation, continued AMTU staff accessibility to medical and appointment records;
* Ability for the AMTU staff to access medical and appointment records for a maximum of 78 weeks after enrollment or through February 2017, whichever occurs first;
* Ability to understand spoken English;
* Willing and able to provide signed informed consent or assent;

NOTE: If consent/assent is obtained > 4 weeks prior to the enrollment date, reaffirmation of consent must be obtained prior to starting the Baseline visit.

-Parent or Legal Guardian permission, if applicable; and

In addition to all the criteria listed above, to be considered eligible for enrollment after August 31, 2015, an individual must also meet the following criterion.

-Must be considered either: (a) newly engaged in HIV medical care defined as no previous initial comprehensive HIV medical care visit with consent occurring before, at the time of, or within four weeks following that initial comprehensive visit; or (b) newly re-engaged in HIV medical care defined as attending the last medical appointment more than 52 weeks ago.

*NOTE: The initial HIV medical care appointment is defined as a routine HIV medical appointment where the adolescent attends with a medical provider authorized to prescribe medication.

This HIV medical appointment must be a non-emergency, routine condition-focused exam AND one or more of the following:

* CD4, VL lab draw and/or review of these lab results;
* Discussion around HIV ART options;
* Primary and/or secondary HIV prevention education and counseling; or
* Diagnosis and treatment of complications of HIV, and of AIDS-defining conditions.

Exclusion Criteria:

* Presence of serious psychiatric symptoms (e.g., active hallucinations, thought disorder) that would impair the individual's ability to provide true informed consent or participate in the baseline ACASI*;
* Visibly distraught (e.g., suicidal, homicidal, exhibiting violent behavior) at the time of consent or the baseline ACASI*; or
* Intoxicated or under the influence of alcohol or other substances at the time of consent or the baseline ACASI*

  * NOTE: If consent/assent is obtained prior to the enrollment date, assessment for these exclusion criteria must be performed again prior to administration of the baseline ACASI (Enrollment). If any are present, the subject cannot be enrolled; do not administer the ACASI. Reassessment of eligibility and enrollment may take place at a later date per the discretion of the treating clinician.

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 1. Behaviorally-infected, HIV-positive adolescents and young adults who are currently receiving or plan to receive their medical care at any clinical site that is part of the AMTU;
  2. Ages 13 through 24, inclusive, at the Baseline visit;
  3. Males and females;
  4. Ability to understand spoken English; and
  5. Ability for the AMTU staff to access the subject's medical records for a maximum of 78 weeks after enrollment or through February 2017, whichever occurs first.
Sampling Method: Non-Probability Sample
Enrollment: 924 (Actual)
Dates: Start 2015-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects engaged in care at Baseline, per subject year, as defined by the HRSA HAB measure | Baseline
The proportion of subjects engaged in care at Week 26, per subject year, as defined by the HRSA HAB measure | Week 26
The proportion of subjects engaged in care at Week 52, per subject year, as defined by the HRSA HAB measure | Week 52
The proportion of subjects engaged in care at Week 78, per subject year, as defined by the HRSA HAB measure | Week 78
The proportion of subjects engaged in care at Baseline, per subject year, as defined by the DHHS measure | Baseline
The proportion of subjects engaged in care at Week 26, per subject year, as defined by the DHHS measure | Week 26
The proportion of subjects engaged in care at Week 52, per subject year, as defined by the DHHS measure | Week 52
The proportion of subjects engaged in care at Week 78, per subject year, as defined by the DHHS measure | Week 78
The proportion of subjects prescribed antiretroviral therapy at Baseline per subject year | Baseline
The proportion of subjects prescribed antiretroviral therapy at Week 26 per subject year | Week 26
The proportion of subjects prescribed antiretroviral therapy at Week 52 per subject year | Week 52
The proportion of subjects prescribed antiretroviral therapy at Week 78 per subject year | Week 78
The proportion of subjects that have achieved viral suppression at Baseline per subject year | Baseline
The proportion of subjects that have achieved viral suppression at Week 26 per subject year | Week 26
The proportion of subjects that have achieved viral suppression at Week 52 per subject year | Week 52
The proportion of subjects that have achieved viral suppression at Week 78 per subject year | Week 78

SECONDARY OUTCOMES:
The proportion of subjects with advanced HIV disease at time of first clinical visit defined as a CD4 count < 200 cells/mm3 | Baseline
The incidence of STIs in the study population as an indicator of transmission risk at Baseline | Baseline
The incidence of STIs in the study population as an indicator of transmission risk at Week 26 | Week 26
The incidence of STIs in the study population as an indicator of transmission risk at Week 52 | Week 52
The incidence of STIs in the study population as an indicator of transmission risk at Week 78 | Week 78
Number of subjects with mental health issues at Baseline | Baseline
Number of subjects engaging in substance use at Baseline | Baseline
Number of subjects engaging in sexual risk behaviors at Baseline | Baseline
ART adherence rate at Baseline | Baseline
Frequency of missed clinic visits at Baseline | Baseline
Frequency of missed clinic visits at Week 26 | Week 26
Frequency of missed clinic visits at Week 52 | Week 52
Frequency of missed clinic visits at Week 78 | Week 78
Types of services available at each AMTU at Baseline | Baseline
Types of services available at each AMTU at 48 weeks after Baseline | Week 48
Types of services available at each AMTU at 96 weeks after Baseline | Week 96
Proportion of subjects notifying their sexual partners after learning their HIV status | Baseline
Timing of subjects notifying their partners after learning about their HIV status | Baseline
Proportion of subjects with whom partner notification was discussed | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bret Rudy, MD, Principal Investigator — NYU Langone Health
Locations (14):
- United States (14):
  - University of Colorado/The Children's Hospital, Aurora, California
  - Children's Hopsital of Los Angeles, Los Angeles, California
  - Children's Hospital National Medical Center, Washington D.C., District of Columbia
  - University of Miami School of Medicine, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Stroger Hospital of Cook County, Chicago, Illinois
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Fenway Institute, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Montefiore Medical Center, The Bronx, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine/Texas Children's Hospital, Houston, Texas

REFERENCES:
- See also: ATN website — http://atnonline.org